CLINICAL TRIAL: NCT02790463
Title: A Novel Centralized 'Virtual' Gout Clinic for Chronic Gout Management (NIAMS :CoRT)
Brief Title: Virtual Gout Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Nebraska (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Jeff Curtis, MD, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X121119002
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Gout
Keywords: Allopurinol
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Participants recruited in this arm will receive their usual care for gout as they normally would
- Intervention (Active Comparator): Participants recruited to this arm will receive their usual gout care + pharmacist-led intervention
  Interventions: Behavioral: Pharmacist-Led Intervention

INTERVENTIONS:
Behavioral: Pharmacist-Led Intervention — Pharmacists will conduct outreach primarily via an automated telephone interactive voice recognition system and direct (telephone) contact
  Arms: Intervention

SUMMARY:
The overarching goal of the investigators project is to identify best practices in gout and hyperuricemia management, translate these evidence-based practices into a highly generalizable strategy for optimal delivery of gout care, and implement and evaluate such a strategy in a large, population-based healthcare setting. With the use of novel but readily-accessible technology, the investigators will examine the use of a novel, large-scale, and relatively low-cost pharmacy-based intervention, with the goal of optimizing urate lower therapy (ULT) in chronic gout treatment.

DETAILED DESCRIPTION:
Gout is a chronic and progressive form of arthritis occurring as a result of monosodium urate deposition in the joints and surrounding tissues. Despite its extremely well known pathogenesis and the availability of highly efficacious therapies, gout continues to lead to considerable morbidity and mortality due to poor management and limited therapeutic adherence. The investigators translational research study will address this deficit in evidence implementation.

The treatment of chronic gout is based primarily on the use of urate lower therapy (ULT) to reduce the frequency of, and eventually eliminate, acute flares in addition to reducing the risk of progressive joint destruction. There are currently four ULT agents approved for the treatment of gout in the United States (US) including probenecid (a uricosuric), pegloticase (a biologic therapy approved for treatment-refractory gout), allopurinol, and febuxostat. Available for more than 40 years, allopurinol remains the most frequently prescribed ULT, accounting for ~99% of all ULT prescriptions. Many early studies confirmed the robust urate lowering effect of allopurinol, a treatment also yielding ample improvements in long-term outcomes including a reduction in gouty flares. A recent 28-week randomized trial examining fixed dose daily allopurinol revealed a 34% reduction in serum urate concentrations vs. a decrease of 3-4% for those receiving placebo. There are factors that contribute to sub-optimal allopurinol administration and likely include, but are not limited to: 1) failure of prescribers to appropriately titrate allopurinol dose to achieve optimal serum urate target levels; 2) poor long term patient adherence to therapy; 3) drug intolerance, recognizing that this affects only a small proportion of patients; 4) limited data regarding the effectiveness of doses exceeding 300 mg/day; and 5) concerns regarding increased toxicity with higher doses, particularly in the context of chronic kidney disease (CKD).

To date, there have been no published studies examining the impact of a large scale intervention implemented to optimize allopurinol administration in gout. Intervention studies that have been done have universally involved small sample sizes and have been limited to single centers, substantially limiting the external validity of these efforts. The impact of these interventions, largely employing prescription audits and performance feedback to providers, have either gone unreported or have been quite modest in effect. Given the potential cost-effectiveness of allopurinol in gout treatment compared to alternative ULTs and the growing number of reports that have consistently characterized its everyday use as sub-optimal, interventions focused on improving and optimizing allopurinol administration in the context of 'real-life' gout care are urgently needed.

ELIGIBILITY:
Inclusion Criteria:

* At least one prior International Classification of Disease (ICD) 9 code for gout (274.xx)
* Received a new prescription for allopurinol, defined as no prior allopurinol prescription in the preceding 12 months

Exclusion Criteria:

* No prior ICD9 code for gout (274.xx)
* Did not receive a new prescription for allopurinol, defined as no prior allopurinol prescription in the preceding 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1463 (Actual)
Dates: Start 2013-01; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Permanente, Pasadena, California

IPD SHARING:
Plan to Share IPD: No
No, not permitted by data use agreements

REFERENCES:
- [Derived] Mikuls TR, Cheetham TC, Levy GD, Rashid N, Kerimian A, Low KJ, Coburn BW, Redden DT, Saag KG, Foster PJ, Chen L, Curtis JR. Adherence and Outcomes with Urate-Lowering Therapy: A Site-Randomized Trial. Am J Med. 2019 Mar;132(3):354-361. doi: 10.1016/j.amjmed.2018.11.011. Epub 2018 Nov 29. PMID 30503879

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 782 | 681
Completed | 782 | 372
Not Completed | 0 | 309

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 782 | 681 | 1463
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (14.4) | 58.6 (14.2) | 58.3 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 134 | 269
  Male | 647 | 547 | 1194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 182 | 175 | 357
  Not Hispanic or Latino | 600 | 506 | 1106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 203 | 135 | 338
  Native Hawaiian or Other Pacific Islander | 38 | 31 | 69
  Black or African American | 109 | 77 | 186
  White | 133 | 127 | 260
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 296 | 308 | 604
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 782 | 681 | 1463
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 31.5 (6.5) | 31.5 (7.6) | 31.5 (7.0)
Serum urate, mean [Mean (Standard Deviation); unit: mg/dl] | 8.4 (1.6) | 8.4 (1.6) | 8.4 (1.6)
Serum creatinine, mean [Mean (Standard Deviation); unit: mg/dl] | 1.16 (.35) | 1.16 (.35) | 1.16 (.35)
Allopurinol dose, mean [Mean (Standard Deviation); unit: mg/day] | 188 (101) | 190 (98) | 189 (100)
Colchicine use [Count of Participants; unit: Participants] | 419 | 375 | 794
Prescription NSAID use [Count of Participants; unit: Participants] | 385 | 350 | 735
Glucocorticoid use [Count of Participants; unit: Participants] | 293 | 251 | 544
Thiazide diuretic [Count of Participants; unit: Participants] | 71 | 80 | 151
Loop diurectic [Count of Participants; unit: Participants] | 68 | 47 | 115
Diabetes mellitus [Count of Participants; unit: Participants] | 170 | 157 | 327
hypertension [Count of Participants; unit: Participants] | 452 | 407 | 859

OUTCOME MEASURES:

1. Primary Outcome: sUA < 6.0 mg/dl at 1 Year
Description: Achievement of serum uric acid (sUA) < 6.0 mg/dl at 1 year
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 782 | 681
Participants | 117 | 204

2. Primary Outcome: Adherence to Medication
Description: Adherence to prescribed medication
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 782 | 681
Participants | 250 | 341

ADVERSE EVENTS:
Time Frame: 2 year study period
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 0/782 | 0/681
Serious Adverse Events (participants affected / at risk) | 1/782 | 1/681
Other Adverse Events (participants affected / at risk) | 0/782 | 0/681
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=782) | Intervention (N=681)
Toxic epidermal necolysis (TENs) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Severe cutaneous reaction
Drug rash with eosinophilia and systemic symptoms (DRESS) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Severe cutaneous reaction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT02790463/Prot_SAP_000.pdf